CLINICAL TRIAL: NCT03710811
Title: Observational Study of Drug Naive Type 2 Diabetes Receiving Continuous Subcutaneous Insulin Infusion Therapy
Brief Title: Observational Study of Drug Naive Diabetes Receiving Insulin Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Dalong Zhu, Doctor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: INSULIN001
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Type 2 Diabetes
Keywords: insulin; drug naive
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample with DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 2 Diabetes: drug naive Type 2 Diabetes received insulin therapy
  Interventions: Drug: Insulin
- normal control: healthy volunteers as normal control

INTERVENTIONS:
Drug: Insulin — Continuous Subcutaneous Insulin Infusion
  Groups: Type 2 Diabetes

SUMMARY:
A multi-centre, open-label trial to investigate the efficacy and possible mechanism of Continuous Subcutaneous Insulin Infusion treatment in patients with drug naive type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

for type 2 diabetes:

1. Male or female age ≧ 25 years and ≦75 years old
2. HbA1c ≧8.0%
3. durg naive

for normal controls：

1. Male or female age ≧ 25 years and ≦75 years old
2. Normal glucose tolerance confirmed by oral glucose tolerance test

Exclusion Criteria:

1. Islet antibody positive
2. Athletes, has a history of skeletal muscle injury ( trauma or surgery ), skeletal muscle wasting diseases ( such as mitochondrial myopathy, muscular atrophy, etc )
3. Acute infection(such as cute upper respiratory infection, acute pneumonia)
4. long-term use of non-steroidal anti-inflammatory drugs, corticosteroids and immunosuppressive drugs
5. consists with other endocrine diseases
6. pregnancy
7. cancer
8. use of antibiotics in 3 months
9. chronic digestive inflammations
10. magnetic resonance imaging contraindications

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: drug naive type 2 diabetes and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Circulating immunity cell profiles | 7 days
  profiles of circulating immunity cells such as T cells

SECONDARY OUTCOMES:
skeletal muscle parameter | 7 days
  skeletal muscle parameters in magnetic resonance imaging

OTHER OUTCOMES:
fasting blood glucose | 7 days
  fasting blood glucose

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - at Division of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu
  - Zhejiang Provincial People'S Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
no plan to share

REFERENCES:
- [Derived] Zhang W, Wang H, Liu F, Ye X, Tang W, Zhang P, Gu T, Zhu D, Bi Y. Effects of Early Intensive Insulin Therapy on Endothelial Progenitor Cells in Patients with Newly Diagnosed Type 2 Diabetes. Diabetes Ther. 2022 Apr;13(4):679-690. doi: 10.1007/s13300-021-01185-w. Epub 2021 Dec 11. PMID 34894328
- [Derived] Tang W, Zhang B, Wang H, Li M, Wang H, Liu F, Zhu D, Bi Y. Improved skeletal muscle energy metabolism relates to the recovery of beta cell function by intensive insulin therapy in drug naive type 2 diabetes. Diabetes Metab Res Rev. 2019 Oct;35(7):e3177. doi: 10.1002/dmrr.3177. Epub 2019 May 27. PMID 31077529